CLINICAL TRIAL: NCT01275456
Title: Validation of an Environmental Exposure Chamber for Inhalation Studies With House Dust Mite Allergen in Patients With Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Prof. Dr. Jens Hohlfeld, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 09/01 Valex1
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Allergy to House Dust Mite
Keywords: allergen provocation; environmental challenge; allergen chamber; house dust mite; immunotherapy
MeSH Terms: conditions — Dust Mite Allergy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Exposure to house dust mite — 0 SQE/qm for 4 hours 250 SQE/qm for 4 hours 500 SQE/qm for 4 hours 1000 SQE/qm for 4 hours

SUMMARY:
This clinical validation study is aimed at testing the efficacy of a new environmental challenge chamber (ECC) to induce symptoms of allergic rhinitis in patients allergic to house dust mite. The symptoms will be recorded on a validated symptom score as Total Nasal Symptom Score (TNSS), allowing for determine whether the challenge is dose dependent and reproducible.

DETAILED DESCRIPTION:
At Fraunhofer ITEM, a novel technique to create an atmosphere loaded with allergenic particles was recently developed. In brief, particles are produced in a combined process of nebulization and drying of a solution containing soluble allergenic extracts and lactose. The particle size distribution is regulated by the droplet size distribution and the lactose concentration in the solution, while the allergen content can be chosen independently. Thus, the Fraunhofer scientists have created a universal tool which provides them with the possibility to create atmospheres containing allergenic particles of arbitrary sizes containing a variety of different allergens. By choosing particle sizes preferentially depositing in the nose (above 10 µm) or the lungs (5 to 10 µm), and selecting allergen concentrations commonly found in the environment, it is possible to build up challenge atmospheres for a large variety of indications.

The first clinical application of this new method will be to create an atmosphere simulating the natural exposure to house dust mite allergens. The challenge aerosol will be composed of lactose as carrier material and the two major allergens Der p1 and Der p2 of house dust mites originating from a licenced allergen extract for inhaled challenge.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18-55 years.
* Non smokers or ex-smokers with a history of less than 10 pack years, having been nonsmokers for at least the last 12 months.
* History of allergic rhinitis to house dust mite. Subjects with mild intermittent asthma that is controlled with occasional use of as-needed short-acting beta-agonists may be included.
* Normal lung function (FEV1 ≥ 80 % pred)
* Positive skin prick test for dermatophagoides pteronyssinus.
* Able and willing to give written informed consent to take part in the study.
* Available to complete all study measurements.
* Women will be considered for inclusion if they are:

  * Not pregnant, as confirmed by pregnancy test (see flow chart) and not nursing.
  * Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).
  * Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).

Exclusion Criteria:

* History of a respiratory tract infection and/or exacerbation of asthma within 4 weeks before the screening.
* Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
* Administration of oral, injectable or dermal corticosteroids within 8 weeks or intranasal and/or inhaled corticosteroids 4 weeks prior to enrollment.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Any structural nasal abnormalities or nasal polyps on examination, history of frequent nose bleeding or recent nasal surgery.
* Conditions or factors, which would make the subject unlikely to be able to stay in the Fraunhofer ECC for four to six hours.
* Specific Immunotherapy (SIT) within the last two years prior to screening.
* Risk of non-compliance with study procedures.
* Participation in another clinical trial 30 days prior to enrolment.
* Any contraindication for adrenalin use (e.g. use of local and systemic beta-blockers)
* Intolerance to any excipients especially lactose and/or milk products
* History of drug or alcohol abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom score (TNSS) | During 4 hours of challenge
  To assess the effect of a 4 hour-environmental allergen challenge with house dust mite extract in an ECC on the total nasal symptom score (TNSS), defined as the sum of obstruction, rhinorrhea, itch, and sneeze, each of which has been scored on a scale from 0 to 3.

SECONDARY OUTCOMES:
Rhinomanometry | During 4 hours of challenge
  To assess the effect of a 4-hour-environmental allergen challenge with house dust mite extract.
visual analogue scale (VAS) for total nasal symptoms | During 4 hours of challenge
  To assess the effect of a 4-hour-environmental allergen challenge with house dust mite extract
Nasal secretion | during 4 hours of challenge
  To assess the effect of a 4-hour-environmental allergen challenge with house dust mite extract.
Exhaled Nitric Oxide (NO) | during and up to 24 hours after challenge
  To assess the effect of a 4-hour-environmental allergen challenge with house dust mite extract.
FEV1 | during and up to 24 hours after challenge
  To assess the effect of a 4-hour-environmental allergen challenge with house dust mite extract.

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer-Institute for Toxicology and Experimental Medicine, Hanover, Germany

REFERENCES:
- See also: Sponsor's homepage — http://www.item.fraunhofer.de